CLINICAL TRIAL: NCT01922570
Title: Economic Investigation of Diarrhoea During Nutritional Support in Intensive Care Unit Patients
Brief Title: Economics of Diarrhoea in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Head, Clinical Nutrition, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAC 07-098
Record Dates: First submitted 2013-06-24; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Critical Illness
Keywords: Enteral nutrition; Supplemental parenteral nutrition; Critical illness; ICU patients; diarrhea
MeSH Terms: conditions — Critical Illness; Diarrhea | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary supplements:parenteral nutrition (Experimental): supplemental parenteral nutrition and enteral nutrition in case of failure (intake below 60% of energy needs) of enteral nutrition by day 3 after admission in the ICU or enteral nutrition only.
  Interventions: Dietary Supplement: nutrition

INTERVENTIONS:
Dietary Supplement: nutrition — comparion of enteral versus enteral and supplemental parenteral nutrition
  Other Names: Enteral+parenteral nutrition

SUMMARY:
Enteral nutrition (EN) is the first choice route for nutritional support in ICU patients with a functioning digestive tract. Nevertheless, EN alone is often associated with digestive intolerance, including diarrhoea. In case of diarrhoea, EN is often reduced or discontinued, resulting in insufficient energy and protein intakes and increase complications rate in ICU patients. Diarrhoea is more frequent in ICU patients receiving EN that in those without EN or on Parenteral nutrition (PN). This difference is likely to be related to the level of EN administration needed to optimize the coverage of nutritional needs at a time when the gut has reduced absorptive capacity. Diarrhoea is suspected to have a negative economic impact on global cost, because the management of patients with diarrhoea is time-consuming for the nurses and all medical staff, it requires investigations (water and electrolytes balances, microbiology investigations, etc.) and treatments (anti-diarrhoeal drugs, antibiotics, etc). However, the economic impact of diarrhoea related to EN or the combination of EN and PN has never been evaluated in the ICU setting.

DETAILED DESCRIPTION:
Rationale: Enteral nutrition (EN) is the first choice route for nutritional support in ICU patients with a functioning digestive tract (1). Nevertheless, EN alone is often associated with digestive intolerance, including diarrhoea (2,3). In case of diarrhoea, EN is often reduced or discontinued, resulting in insufficient energy and protein intakes (4) and increase complications rate in ICU patients (5-7). Diarrhoea is more frequent in ICU patients receiving EN that in those without EN or on PN. This difference is likely to be related to the level of EN administration needed to optimize the coverage of nutritional needs at a time when the gut has reduced absorptive capacity. Diarrhoea is suspected to have a negative economic impact on global cost, because the management of patients with diarrhoea is time-consuming for the nurses and all medical staff, it requires investigations (water and electrolytes balances, microbiology investigations, etc.) and treatments (anti-diarrhoeal drugs, antibiotics, etc). However, the economic impact of diarrhoea related to EN or the combination of EN and PN has never been evaluated in the ICU setting.

Hypothesis: We made the hypothesis that the extra cost related to the combination of EN and PN prescription is compensated by the decrease in cost secondary to a reduced prevalence of EN-related diarrhoea, which means that the combination of EN and PN is cost-efficient strategy for optimal feeding in ICU patients.

It is known that:

* diarrhoea is more frequent in ICU patients with EN than in those without EN,
* the higher the EN delivery rate, the higher the risk of diarrhoea,
* the combination of EN and PN decreases the need for high EN delivery rate to fully cover the patients' nutritional needs.

It is likely that:

* diarrhoea-related care costs of EN are higher than those observed in patients receiving a combination of EN and PN,
* extra costs related to the combination of EN and PN prescription are compensated by the decrease in costs secondary to a reduced prevalence of EN-related diarrhoe,

Study objectives:

* To determine retrospectively the global prevalence of diarrhoea in all the ICU patients during a three month period.
* To determine prospectively the prevalence of diarrhoea in the ICU patients included in the "SPN study" on EN alone or EN + PN. To validate this current prevalence of diarrhoea by comparison to the retrospective prevalence rate in our ICU.
* To determine prospectively the diarrhoea-related overall costs in the patients of the "SPN study" on EN alone or EN + PN.

Study endpoints: Three categories of study endpoints will be assessed: economic, gastrointestinal tolerance, feeding protocol.

* Economic in Swiss francs:

  * Nursing time for the management of diarrhoea (changes of bed-clothes and disposable nappies)and of nutritional support (time spent to prepare and administer EN and/or PN solutions, introduction and maintenance of naso-gastric tube, catheters, lines, etc)
  * Medical time for prescriptions in seconds of the investigations required by the managment of diarrhoea and of the material costs: drugs (antibiotics, drugs inhibiting motility, etc.), bed-clothes, gloves, disposable nappy, EN and/or PN solutions.
* Gastrointestinal tolerance: Symptoms such as as diarrhoea, defined as liquid stools, defined as three or more liquid stools per day, for at least 1 day, and nausea, vomiting, diarrhoea, flatulence, or constipation.
* Feeding protocol: the route of feeding (EN versus PN), the type, quantities and modalities for delivering nutrition products.
* Inclusion criteria: All patients already included in the "SPN study" receiving.
* Exclusion criteria: none.
* Risk and benefit: The present study will not induce any change to the cares defined in the "SPN study" protocol.
* Additional data recorded to the "SPN study" database:

Clinical data: Diarrhoea: number and frequency of stools for the 5 intervention days (Day 3 and 8) and digestive tolerance: measurements of gastric residues according to ou on-going ICU protocol, frequency of nausea, vomiting, flatulence and constipation.

Economic data: Time measurements for physicians activities using a chronometer:Management of nutritional support, Prescription of nutritional support and micronutrients, Investigations related to the management of nutritional support: upper gastrointestinal endoscopy for the insertion of nasojejunal or nasogastric feeding tube or for the investigation of digestive intolerance, Insertion of central venous catheter, Prescription of drugs for the management of diarrhoea: antibiotics, drugs inhibiting motility, etc., Prescription of investigations for the management of diarrhoea: lower gastrointestinal endoscopy, microbiology for the analysis of stools, blood analysis (electrolytes, renal fucntion, etc)

The cost for each item will be calculated according to the cost of manpower based on mean Swiss data as previously described (8).

- Time measurements for nurses activities using a chronometer:

* Management of nutritional support

  * Preparation of nutritional support: installation of pumps, connections of bottles with bags, addition of micronutrients (vitamins and trace elements) and insertion of naso-gastric tube for EN
  * Monitoring: calculation and setting of flow rates
  * Supervision: noting all observations regarding nutritional support in patient nursing file, changes of bottles and bags
* Management of diarrhoea

  * Preparation of anti-diarrhoea drugs or antibiotics
  * Nursing cares: cleaning, resetting of bed-clothes, wearing of disposable nappies, wound-dressings The cost for each item will be calculated according to the cost of manpower based on mean Swiss data as previously described (8).
* Material costs

  * Drugs: antibiotics, anti-diarrhoea drugs
  * Nutritional support: central venous catheters, naso-gastric tubes, cost of one day IV pump utilization, cost of nutrient solutions, additive materials
  * Cleaning and disinfections: bed-clothes, gloves, caps, disposable nappy
  * Statistics:

All patients included in the "SPN study" (9) will provide prospective data about the association between the type of nutritional support (EN, combination of EN and PN) and the occurrence of diarrhoea. We plan to complete this analysis by measuring the economic criteria, as described in the paragraph 7 above. These data will allow to develop an economic model to be applied to all the data acquired in the SPN study.

* Ethics This study protocol is the addendum no 1 to our existing protocol and which is in full compliance with our institution guidelines. Briefly, this extension of the protocol has been approved by the Chief of the ICU before the procedure has been initiated.
* References

  1. Kreymann KG, Berger MM, Deutz NE, Hiesmayr M, Jolliet P, Kazandjiev G, et al. ESPEN Guidelines on Enteral Nutrition: Intensive care. Clin Nutr 2006;25(2):210-23
  2. Homann NH, Kemen M, Fuessenich C, Senkal M, Zumtobel V. Reduction in diarrhea incidence by solute fiber in patients receiving total or supplemental enteral nutrition. J Parenter Enteral Nutr 1994;18:486-90
  3. Rushdi TA, Pichard C, Khater YH. Control of diarrhea by fiber-enriched diet in ICU patients on enteral nutrition: a prospective randomized controlled trial. Clin Nutr 2004;23:1344-1352
  4. Genton L, Dupertuis YM, Romand JA, Simonet ML, Jolliet P, Huber O, et al. Higher calorie prescription improves nutrient delivery during the first 5 days of enteral nutrition. Clin Nutr 2004; 23(3):307-15
  5. Villet S, Chiolero RL, Bollmann MD, Revelly JP, Cayeux RNM, Delarue J, et al. Negative impact of hypocaloric feeding and energy balance on clinical outcome in ICU patients. Clin Nutr 2005;24(4):502-9
  6. Ibrahim EH, Mehringer L, Prentice D, Sherman G, Schaiff R, Fraser V, et al. Early versus late enteral feeding of mechanically ventilated patients: results of a clinical trial. JPEN J Parenter Enteral Nutr 2002;26(3):174-81
  7. Artinian V, Krayem H, DiGiovine B. Effects of early enteral feeding on the outcome of critically ill mechanically ventilated medical patients. Chest 2006;129(4):960-7
  8. Pichard C, Schwarz G, Frei A, Kyle U, Jolliet P, Morel P, Romand JA, Sierro C. Economic investigation of the use of three-compartment total parenteral nutrition bag: prospective randomized unblinded controlled study. Clin Nutr 2000;19:245-251
  9. Heidegger CP, Berger MM, Graf S, et al. (2013). Optimization of energy provision with supplemental parenteral nutrition (SPN) improves the clinical outcome of critically ill patients : a randomized controlled trial. Lancet 381: 385-393

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication to receive enteral nutrition

Exclusion Criteria:

* patients with a contraindication to receive enteral nutrition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cost of diarrhea | day 28
  Swiss francs: All costs (manpower, investigations, treatments) related to diarrhea during the ICU stay up to 28 days are reported as Swiss francs

SECONDARY OUTCOMES:
Use of enteral nutrition | day 28
  The use of enteral nutrition during the ICU stay and its association with the occurence of diarrhea will recorded

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service of Intensive Care, Geneva, Switzerland

REFERENCES:
- [Derived] Heidegger CP, Graf S, Perneger T, Genton L, Oshima T, Pichard C. The burden of diarrhea in the intensive care unit (ICU-BD). A survey and observational study of the caregivers' opinions and workload. Int J Nurs Stud. 2016 Jul;59:163-8. doi: 10.1016/j.ijnurstu.2016.04.005. Epub 2016 Apr 20. PMID 27222461